CLINICAL TRIAL: NCT05760170
Title: An Observational Study to Determine Experience Patterns in Participants of Lung Cancer Clinical Trials
Brief Title: Determining Clinical Trial Experiences of Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81893664
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This trial will admit a wide range of data on the clinical trial experience of lung cancer patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with lung cancer
* Patient has self-identified as planning to enroll in an observational clinical trial
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Pregnant or nursing patients
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients who are actively considering participating in a clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of lung cancer patients who decide to enroll in a clinical trial | 3 months
Rate of patients who remain in a lung cancer clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Menis J, Besse B, Lacombe D. Methodology of clinical trials in lung cancer. Chin Clin Oncol. 2015 Dec;4(4):44. doi: 10.3978/j.issn.2304-3865.2015.11.03. PMID 26730756
- [Background] Schulkes KJ, Nguyen C, van den Bos F, van Elden LJ, Hamaker ME. Selection of Patients in Ongoing Clinical Trials on Lung Cancer. Lung. 2016 Dec;194(6):967-974. doi: 10.1007/s00408-016-9943-7. Epub 2016 Sep 20. PMID 27650509
- [Background] Schulkes KJ, Nguyen C, van den Bos F, Hamaker ME, van Elden LJ. Patient-Centered Outcome Measures in Lung Cancer Trials. Lung. 2016 Aug;194(4):647-52. doi: 10.1007/s00408-016-9903-2. Epub 2016 Jun 10. PMID 27287676

DOCUMENTS (1):
  • Informed Consent Form (2023-02-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT05760170/ICF_000.pdf